CLINICAL TRIAL: NCT01825616
Title: Influence of 6-weeks Supplementation With Vitamin D Portobello Mushroom Powder on Muscle Function and Performance, Innate Immune Function, and Exercise-induced Muscle Damage and DOMS in NASCAR Pit Crew Members
Brief Title: Vitamin D2, Muscle Damage, NASCAR Pitcrew
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Collaborators: Dole Food Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 12_0355
Record Dates: First submitted 2013-04-03; First posted 2013-04-05 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Muscle Function; Muscle Soreness; Vitamin D Status
Keywords: Strength; Anaerobic power; Muscle soreness; Immune function
MeSH Terms: conditions — Myalgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D2 mushroom powder (Experimental): 4000 IU/day vitamin D2 mushroom powder
  Interventions: Dietary Supplement: Vitamin D2 mushroom powder
- Placebo (Placebo Comparator): Mushroom powder without vitamin D2 (not exposed to UV radiation)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D2 mushroom powder — Subjects will be given Portobello mushroom powder with or without vitamin D mixed in soymilk powder in six plastic containers (one for each week of the study). Subjects will ingest one level teaspoon of the product each day (with or without 4,000 IU vitamin D2) and consume during breakfast in one of the following ways: mixed in water, juice, yogurt, or milk.
  Other Names: UV radiated Portobello mushroom powder
  Arms: Vitamin D2 mushroom powder
Other: Placebo — Mushroom powder without vitamin D2
  Arms: Placebo

SUMMARY:
Hypothesis: Six weeks of supplementation with vitamin D (4000 IU/day) using Dole's Vitamin D Portobello Mushroom Powder will increase winter serum vitamin D levels, and improve muscle function and strength, and innate immunity (granulocyte/monocyte phagocytosis and oxidative burst activity), and attenuate exercise-induced muscle damage and DOMS.

DETAILED DESCRIPTION:
Vitamin D2 is found naturally in sun-exposed mushrooms, and vitamin D3 is synthesized in the skin when exposed to sunlight and is present in oil-rich fish such as salmon, mackerel, and herring. Mushrooms contain very little or any vitamin D2 but are abundant in ergosterol, which can be converted into vitamin D2 by ultraviolet (UV) illumination (Eur J Clin Nutr. 2011;65:965-71).

In recent decades, there has been increased awareness of the impact of vitamin D on muscle function (Scand J Med Sci Sports. 2010;20:182-90). In the early 20th century, athletes and coaches felt that ultraviolet rays had a positive impact on athletic performance, and evidence is accumulating to support this view. Both cross-sectional and longitudinal studies support a functional role for vitamin D in muscle, and the discovery of the vitamin D receptor in muscle tissue provides a mechanistic pathway for understanding the role of vitamin D within muscle. Studies in athletes have found that vitamin D status is variable and is dependent on outdoor training time (during peak sunlight), skin color, and geographic location (Pediatr Clin North Am. 2010;57:849-61).

25(OH)D is the best indicator and major form of vitamin D in the blood, with a circulating half-life of 2-3 weeks. Vitamin D deficiency is defined as a plasma vitamin D [25(OH)D] level of less than 20 ng/ml, with vitamin D insufficiency defined as 21-29 ng/ml. Estimates are that 20-100% of children, young and middle-aged adults, and community-dwelling elderly men and women are vitamin D deficient (J Clin Endocrinol Metab. 2011;96:1911-30).

Purpose: To determine if 6 weeks supplementation with Dole Vitamin D Portobello Mushroom Powder (4,000 IU/day) can, 1) increase winter serum vitamin D levels, and measure whether vitamin D supplementation 2) has a chronic influence on muscle function and strength, and innate immune function, and 3) can attenuate exercise-induced muscle damage and delayed onset of muscle soreness (DOMS) in athletes.

ELIGIBILITY:
Inclusion Criteria:

* NASCAR pit crew members
* Willing to avoid food and supplement sources (during the 6-week supplementation period) that are high in vitamin D (specifically canned fish, cod liver oil, salmon, and supplements with high-dose vitamin D).
* Agree to train normally.
* Avoid the use of large dose vitamin/mineral supplements (above 100% recommended dietary allowances), and medications known to affect immune function.
* Avoid the use of tanning beds.
* Willing to adhere to all aspects of the study design.

Exclusion Criteria:

* Not allergic to mushrooms.
* Do not have a heart problem or have been told by your doctor not to engage in vigorous exercise.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2012-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Muscle damage | 6 weeks
  myoglobin (ug/L) and creatine kinase (IU/L) after eccentric resistance exercise
Muscle Function | 6 weeks
  Bench press of body weight, reps to fatigue Vertical jump (watts( 300 yard shuttle run (seconds) 30-sec Wingate anaerobic power test (watts/kg)

SECONDARY OUTCOMES:
Serum vitamin D concentration | 6 weeks
  25(OH)D2 and 25(OH)D3
Immune Function | 6 weeks
  White blood cell differential Myeloperoxidase Immune cell cytotoxicity

CONTACTS AND LOCATIONS:
Overall Officials: David C Nieman, DrPH, Principal Investigator — Appalachian State University
Locations (3):
- United States (3):
  - ASU Human Performance Laboratory, North Carolina Research Campus, Kannapolis, North Carolina
  - ASU-NCRC Human Performance Laboratory, Kannapolis, North Carolina
  - ASU-NCRC Human Performance Lab, Kannapolis, North Carolina

REFERENCES:
- See also: Lab web site — http://www.ncrc.appstate.edu